CLINICAL TRIAL: NCT03787095
Title: Safety and Immunotherapeutic Activity of an Anti-PD-1 Antibody (Cemiplimab) in Participants With HIV-1 on Suppressive cART: A Phase I/II, Double-blind, Placebo-controlled, Ascending Multiple Dose Study
Brief Title: Safety and Immunotherapeutic Activity of an Anti-PD-1 Antibody (Cemiplimab) in Participants With HIV-1 on Suppressive cART
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Stopped by monitoring committee recommendation due to adverse events
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5370; 38399 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — cemiplimab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Cemiplimab (Experimental): Participants received 0.3 mg/kg of cemiplimab, administered at Day 0 and Week 6 for a total of two infusions.
  Participants continued their current non-study provided ART regimen.
  Interventions: Biological: Cemiplimab
- Cohort 1: Placebo (Placebo Comparator): Participants received placebo, administered at Day 0 and Week 6 for a total of two infusions.
  Participants continued their current non-study provided ART regimen.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Cemiplimab — Administered as an intravenous (IV) infusion
  Other Names: REGN2810
  Arms: Cohort 1: Cemiplimab
Biological: Placebo — Diluent for REGN2810, administered as an IV infusion
  Arms: Cohort 1: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety and immunotherapeutic activity of an anti-PD-1 antibody (cemiplimab) in participants with HIV-1 on suppressive combination antiretroviral therapy (cART).

DETAILED DESCRIPTION:
This study evaluated the safety and immunotherapeutic activity of an anti-PD-1 antibody (cemiplimab) in participants with HIV-1 on combination antiretroviral therapy (cART) who have plasma less than the quantification limit of an FDA-approved assay and CD4+ T cell counts ≥350/mm^3.

Participants were planned to be enrolled into three sequential dose-rising cohorts. Participants in each cohort received infusions of either cemiplimab or placebo, with planned administration at study entry (Day 0) and Week 6, for a total of two infusions. All participants continued their non-study provided ART regimen. Enrollment in the second and third cohorts would only open after all participants in the previous cohort had reached week 12 and an evaluation of safety outcomes established that it is safe to dose escalate.

Participants had screening and pre-entry visits and attended study visits on Day 0 and Weeks 1, 2, 4, 6, 7, 8, 10, 12, 16, 20, 24, 28, 36, and 48. Participants were followed for 48 weeks.

Due to observed adverse events which were deemed possibly related to study treatment in two of four treated participants, the study was terminated and did not enroll further participants. The two participants who had adverse events did not receive the second infusion. The treated participants were followed for the planned 48 weeks, while the placebo participant was not followed after a final study visit at week 7.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* On ART for at least 24 months
* Receiving ART with no changes of the components of ART medications within 90 days prior to study entry

  * Changes within drug class, in drug formulation or dose are allowed more than 30 days prior to study entry.
* CD4+ T cell count ≥350 cells/mm^3
* At least two plasma HIV-1 RNA less than the quantification limit of an FDA-approved assay within 18 months

  * A single detectable HIV-1 RNA but less than 1000 copies/mL is allowed if followed by HIV-1 RNA below quantifiable limits.
* HIV-1 RNA level less than the quantification limit of an FDA-approved assay within 90 days prior to study entry
* The following laboratory values within 90 days prior to entry:

  * Absolute neutrophil count (ANC) ≥1500 cells/mm^3
  * Hemoglobin ≥14.0 g/dL for men and ≥12.0 g/dL for women
  * Platelet count ≥150,000/mm^3
  * Creatinine clearance ≥60 mL/min
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal limits
  * Normal thyroid, adrenal and diabetes testing
* Negative tuberculosis (TB) test result, OR documentation of completed TB prophylaxis treatment
* HCV antibody negative result or, if HCV antibody positive, undetectable HCV RNA result
* Negative HBsAg result
* Ability and willingness to provide informed consent.
* Ability and willingness to continue non-study-provided cART throughout the study.
* Female participants must have a negative pregnancy test. Agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization, egg donation) during the study.
* When participating in sexual activity that could lead to pregnancy, agree to use at least two reliable forms of contraception simultaneously during the study through week 48.
* Participants who are not of reproductive potential (women who have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy and/or bilateral oophorectomy or salpingectomy or men who have documented azoospermia or undergone vasectomy) are eligible without requiring the use of contraceptives.
* Weight ≥50 kg (110 pounds)

Exclusion Criteria:

* History of malignancy within the last 5 years.

  * Prior non-melanoma skin cancer (e.g., basal cell carcinoma or squamous cell skin cancer) is not exclusionary with documentation of complete resection at least 3 months prior to enrollment.
* HIV-related opportunistic infections within the last 5 years
* Chronic obstructive pulmonary disease (COPD).
* Prior radiation therapy.
* Active or previously treated active TB.
* Active asthma requiring any treatment in the prior 2 years
* Type I or type II diabetes mellitus.
* History of or active autoimmune disorders including but not limited to inflammatory bowel diseases, scleroderma, severe psoriasis, myocarditis, uveitis, pneumonitis, systemic lupus erythematosus, rheumatoid arthritis, optic neuritis, myasthenia gravis, adrenal insufficiency, hypothyroidism and/or hyperthyroidism, autoimmune thyroiditis, hypophysitis, or sarcoidosis.
* Immune deficiency other than that caused by HIV infection.
* Currently breastfeeding or pregnant.
* Known allergy/sensitivity or any hypersensitivity to mAb-based biologics, cemiplimab (anti-PD-1) or its formulation.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Receipt of investigational drug or use of investigational medical device within 6 months prior to study entry.
* Use of or intent to use immunomodulators (e.g., interleukins, interferons, cyclosporine, systemic corticosteroids exceeding physiologic doses), HIV vaccine, or systemic cytotoxic chemotherapy within 60 days prior to study entry.

  * NOTE: Participants receiving stable physiologic glucocorticoid doses, defined as prednisone ≤10 mg/day or the equivalent, will not be excluded. Stable physiologic glucocorticoid doses should not be discontinued for the duration of the study. In addition, participants receiving topical corticosteroids will not be excluded.
* Any vaccination within 30 days
* HCV treatment within 6 months
* Prior immunoglobulin (IgG) therapy.
* Current use or intent to use biotin ≥5 mg/day, including within dietary supplements.
* History of chronic congestive heart failure or other significant cardiac conditions.
* Any active, clinically significant medical condition that, in the opinion of the site investigator, would place the participant at increased risk.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Gay, MD, Study Chair — Chapel Hill CRS; W. David Hardy, MD, Study Chair — Johns Hopkins University
Locations (3):
- United States (3):
  - Alabama CRS, Birmingham, Alabama
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Chapel Hill CRS, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at:https://submit.mis.s-3.net/ Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.
URL: https://submit.mis.s-3.net/

REFERENCES:
- [Result] Gay CL, Bosch RJ, McKhann A, Moseley KF, Wimbish CL, Hendrickx SM, Messer M, Furlong M, Campbell DM, Jennings C, Benson C, Overton ET, Macatangay BJC, Kuritzkes DR, Miller E, Tressler R, Eron JJ, Hardy WD; A5370 Team. Suspected Immune-Related Adverse Events With an Anti-PD-1 Inhibitor in Otherwise Healthy People With HIV. J Acquir Immune Defic Syndr. 2021 Aug 15;87(5):e234-e236. doi: 10.1097/QAI.0000000000002716. No abstract available. PMID 33929394
- [Derived] Gay CL, Bosch RJ, McKhann A, Cha R, Morse GD, Wimbish CL, Campbell DM, Moseley KF, Hendrickx S, Messer M, Benson CA, Overton ET, Paccaly A, Jankovic V, Miller E, Tressler R, Li JZ, Kuritzkes DR, Macatangay BJC, Eron JJ, Hardy WD; A5370 Team. Safety and Immune Responses Following Anti-PD-1 Monoclonal Antibody Infusions in Healthy Persons With Human Immunodeficiency Virus on Antiretroviral Therapy. Open Forum Infect Dis. 2024 Jan 11;11(3):ofad694. doi: 10.1093/ofid/ofad694. eCollection 2024 Mar. PMID 38449916
- See also: Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids
- See also: National Cancer Institute's (NCI) Common Terminology Criteria for AEs (CTCAE), Version 5.0 — https://ctep.cancer.gov/protocolDevelopment/electronic_applications/docs/CTCAE_v5_Quick_Reference_5x7.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled in August 2019. The final participant was enrolled in September 2019. The study was paused to accrual for emergency review by the study monitoring committee (SMC) in October 2019, followed by the decision to close the study later that month. Participants were recruited from 3 sites in the US.
Groups:
- Cohort 1: Cemiplimab: Participants received 0.3 mg/kg of cemiplimab, with planned administration at Day 0 and Week 6 for a total of two infusions.
  Participants continued their current non-study provided ART regimen.
  Cemiplimab: Administered as an intravenous (IV) infusion
- Cohort 1: Placebo: Participants received placebo, with planned administration at Day 0 and Week 6 for a total of two infusions.
  Participants continued their current non-study provided ART regimen.
  Placebo: Diluent for REGN2810 , administered as an IV infusion
Period: Overall Study
Arm/Group | Cohort 1: Cemiplimab | Cohort 1: Placebo
Started | 4 | 1
Completed | 4 | 1 (Participant had final visit at study week 7 in accordance with decision from team after the study was closed.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Cemiplimab | Cohort 1: Placebo | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [39 to 54] | 52 [52 to 52] | 51 [50 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 0 | 4
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5
CD4 Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 1151 [720 to 1674] | 348 [348 to 348] | 911 [528 to 1391]
CD8 Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 1516 [1188 to 1872] | 286 [286 to 286] | 1508 [867 to 1524]
CD4/CD8 ratio [Median (Inter-Quartile Range); unit: ratio] | 0.90 [0.62 to 0.98] | 1.22 [1.22 to 1.22] | 0.91 [0.88 to 1.05]
HIV-1 RNA [Number; unit: participants]
  <40 copies/mL | 4 | 1 | 5
  >=40 copies/mL | 0 | 0 | 0
Weight [Median (Inter-Quartile Range); unit: kilograms] | 88.8 [77.3 to 98.3] | 101.0 [101.0 to 101.0] | 90.7 [86.9 to 101.0]

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With a Grade >=3 Adverse Event (AE) or Grade >=1 Immune-related AE (irAE) Related to Study Treatment
Description: Relationship to study treatment was judged by the Clinical Management Committee (CMC), blinded to treatment arm. Immune-related AEs include, but were not limited to, pneumonitis, colitis, adrenal insufficiency, or hypothyroidism.
  Adverse events were graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017. Infusion reactions, adrenal insufficiency, and pneumonitis were graded per the National Cancer Institute's (NCI) Common Terminology Criteria for AEs (CTCAE), Version 5.0 guidelines
Time Frame: Study Entry through Week 48 or premature discontinuation
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Cemiplimab | Cohort 1: Placebo
Number analyzed (Participants) | 4 | 1
Participants | 2 | 0

2. Primary Outcome: Count of Participants With a Grade >=1 irAE Related to Study Treatment
Description: as for outcome 1
Time Frame: Study Entry through Week 48 or premature discontinuation
Population: All participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Cemiplimab | Cohort 1: Placebo
Number analyzed (Participants) | 4 | 1
Participants | 2 | 0

3. Secondary Outcome: Change in HIV-1 Gag-specific CD8+ T Cells by Intracellular Staining for CD107a and Interferon Gamma (IFNg) From Baseline to Post-baseline
Description: Change evaluated from baseline (average of pre-entry and entry measures) to post-baseline (average of weeks 2-12 measures). Results for each week are calculated by subtracting the corresponding background control value. If the result was less than zero after background subtraction, the result was set to zero.
Time Frame: Baseline through Week 12
Population: All participants
Measure: Mean (Standard Deviation); unit: Percentage of T cells
Arm/Group | Cohort 1: Cemiplimab | Cohort 1: Placebo
Number analyzed (Participants) | 4 | 1
Percentage of T cells | 0.01 (0.07) | 0.09 (NA) — No standard deviation due to N=1
Statistical Analysis 1: Comparison: Cohort 1: Cemiplimab; Null hypothesis: There is no change from baseline to post-baseline among participants treated with Cemiplimab. Per the analysis plan, only participants in the Cemiplimab arm are evaluated; Test type: Superiority; p = 0.71, t-test, 2 sided

4. Secondary Outcome: Change in HIV-1 Gag-specific CD8+ T Cells by Intracellular Staining for IFNg or CD107a Alone From Baseline to Post-baseline
Description: as for outcome 3
Time Frame: Baseline through Week 12
Population: All participants
Measure: Mean (Standard Deviation); unit: Percentage of T cells
Arm/Group | Cohort 1: Cemiplimab | Cohort 1: Placebo
Number analyzed (Participants) | 4 | 1
Percentage of T cells | 0.00 (0.70) | 2.52 (NA) — No standard deviation due to N=1
Statistical Analysis 1: Comparison: Cohort 1: Cemiplimab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 1.00, t-test, 2 sided

5. Secondary Outcome: Change in Polyfunctional Response of HIV-1 Gag-specific CD8+ T Cells by Intracellular Staining for IFNg, CD107a, IL-2, and Tumor Necrosis Factor Alpha (TNFa) From Baseline to Post-baseline
Description: Change evaluated from baseline (average of pre-entry and entry measures) to post-baseline (average of weeks 2-12 measures). Polyfunctional response was defined as being positive for two or more cytokines. Results for each week are calculated by subtracting the corresponding background control value. If the result was less than zero after background subtraction, the result was set to zero.
Time Frame: Baseline through Week 12
Population: All participants
Measure: Mean (Standard Deviation); unit: Percentage of T cells
Arm/Group | Cohort 1: Cemiplimab | Cohort 1: Placebo
Number analyzed (Participants) | 4 | 1
Percentage of T cells | 0.24 (0.42) | -0.86 (NA) — No standard deviation due to N=1
Statistical Analysis 1: Comparison: Cohort 1: Cemiplimab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.33, t-test, 2 sided

6. Secondary Outcome: Change in HIV-1 Gag-specific CD8+ T Cells by Intracellular Staining for IFNg and CD107a After Each Infusion
Description: Change evaluated from baseline (average of pre-entry and entry measures) to after the first dose (average of Weeks 2-6), and from baseline to after the second dose (average of Weeks 8-12). Results for each week are calculated by subtracting the corresponding background control value. If the result was less than zero after background subtraction, the result was set to zero.
Time Frame: Baseline through Week 12
Population: As per the analysis plan, only participants who received two study treatment infusions (at baseline and week 6) of the study treatment Cemiplimab are included (therefore the Placebo arm is not listed). The two participants with adverse events only received one infusion at baseline and are not included.
Measure: Mean (Standard Deviation); unit: Percentage of T cells
Arm/Group | Cohort 1: Cemiplimab
Number analyzed (Participants) | 2
Percentage of T cells
  After first dose | -0.01 (0.02)
  After second dose | 0.05 (0.20)

ADVERSE EVENTS:
Time Frame: Study entry through week 48 or premature discontinuation.
Description: AEs were defined as using the following criteria: All Grade ≥1 AEs, all suspected or confirmed irAEs, all infusion reactions, all AEs that led to a change in study intervention, all AEs meeting SAE definition or Expedited Adverse Event (EAE) reporting requirement, and all targeted events as specified in the protocol.
  The DAIDS AE Grading Table, V2.1 was used. Infusion reactions, adrenal insufficiency, and pneumonitis were graded by CTCAE guidelines, v5.0.
Arm/Group | Cohort 1: Cemiplimab | Cohort 1: Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/1
Other Adverse Events (participants affected / at risk) | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Cemiplimab (N=4) | Cohort 1: Placebo (N=1)
Thyroiditis (Endocrine disorders) | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0
Thyroxine increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Cemiplimab (N=4) | Cohort 1: Placebo (N=1)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood bicarbonate decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to adverse events and was not able to fully evaluate the efficacy outcomes due to the small number of accrued participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (3):
  • Study Protocol (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT03787095/Prot_001.pdf
  • Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT03787095/SAP_002.pdf
  • Informed Consent Form (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT03787095/ICF_000.pdf